CLINICAL TRIAL: NCT03744195
Title: Effect of Kinesotaping on Management of Supraspinatus Tendinitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RiphahtMahnoor Anwar
Record Dates: First submitted 2018-11-14; First posted 2018-11-16 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Supraspinatus Tendinitis
Keywords: Supraspinatus; Tendinitis; Kinesotaping
MeSH Terms: conditions — Tendinopathy

STUDY DESIGN:
Intervention Model Description: Experimental study
Who Masked: Investigator
Masking Description: This will be a single blinded study.Participants will be randomly allocated to Group (I)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I Experimental Kinesotaping (Experimental): Application of kinesotaping along with conventional treatment
  Interventions: Other: Group I Experimental Kinesotaping
- Group II conventional training group (Active Comparator): Application of conventional treatment
  Interventions: Other: Group II conventional training group

INTERVENTIONS:
Other: Group I Experimental Kinesotaping — For application of kinesotaping following procedure will be adopted:
  1. The skin will be cleaned properly with alcohol
  2. The first strip will be applied in Y-shape (15-20% stretch) surrounding the deltoid muscle to provide inhibition and muscle relaxation
  3. A second strip (I-shape) will be applied for functional correction (50-75% stretch), passing over the supraspinatus, trapezius, glenohumeral joint and middle deltoid Daily Strengthening Exercises (3 sets / 10~30 reps) Joint mobilization (3 sets / 60 seconds hold / 30 seconds interval) Stretching Exercises (3 sets / 30 seconds hold / 30 seconds interval
  Arms: Group I Experimental Kinesotaping
Other: Group II conventional training group — Joint mobilization (3 sets / 60 seconds hold / 30 seconds interval) Stretching Exercises (3 sets / 30 seconds hold / 30 seconds interval) Strengthening Exercises (3 sets / 10~30 reps)
  Arms: Group II conventional training group

SUMMARY:
Supraspinatus tendonitis is a common clinical problem that causes functional and labor disabilities. It is the most frequent cause of shoulder pain. Manual therapy is a common intervention used by physical therapist for management of supraspinatus tendonitis. Joint mobilization, stretching and strengthening exercises are commonly used techniques for management of this condition. In this study KT will be added to conventional manual therapy and its efficacy will be investigated.

The study design will be Randomized Clinical Trial (RCT) that will be used to compare the effects of KT added to manual therapy for management of supraspinatus tendonitis. 38 patients will be participate in this study who will be assigned randomly (biased coin method) to experimental and control groups (19+19). The data collection will be carried out at Railway Hospital Rawalpindi. Patients with shoulder pain at rest and positive for special tests (Neer's, Empty Can, Drop Arm, Hawkin's Kennedy) will be included in this study. There is no restriction on gender and age group will be between 25 and 60 years. Patients with cervical post op, referred pain, open wounds, allergic to KT and with signs of radiculopathy will be excluded from this study. Pre and post treatment evaluation will be done using Visual Analog Scale (VAS), Shoulder Pain and Disability Index (SPADI) and goniometry. Data will be collected on 1st day, 4th day and 7th day for both groups. After data collection is completed, SPSS will be used to analyze the collected data

DETAILED DESCRIPTION:
Shoulder pain is a very common musculoskeletal disorder affecting a large portion of population . Prevalence ranges from 6% to 26% and it is estimated that 33% of population will have one episode of shoulder pain in lifetime. Rotator cuff tendonitis is considered as most common pathology of shoulder . Supraspinatus is one of the four muscles that can cause rotator cuff tendonitis. It is a common clinical disorder that causes functional and labor disorders. It is also the most frequent cause of shoulder pain.

The origin of supraspinatus is fossa of scapula and its insertion is at superior facet on greater tuberosity of humerus. The nerve supply is at C4, C5 and C6. The main function of supraspinatus is abduction of shoulder.

Indications: Supraspinatus tendonitis present following conditions

1. Pain and inflammation
2. Decreased ROM
3. Decreased strength
4. Decreased functional activity Injury Mechanisms: Supraspinatus tendonitis is caused by extrinsic as well as intrinsic factors. Extrinsic factors include increased subacromial activity, trauma, overhead activity, soft tissue imbalance, eccentric muscle overload and glenohumeral laxity. Intrinsic factorare acromial morphology, aging, acromioclavicular arthrosis and coracoacromial ligament hypertrophy.

Kinesiotaping (KT) is widely used in clinical settings for rehabilitation of shoulder disorders . It is designed to facilitate the body's natural healing process while providing support and stability to muscles and joints without restricting the body's range of motion. The functioning of kinesio tap is based on following:

1. Lifting effects of epidermis layers and papillary dermis, caused by micro-convolutions formed on the taped skin .
2. Due to wrinkles generated by the KT, vascular networks in deep vessels under the skin are increased, reducing swelling and inflammation in injured tissues .
3. KT contributes to pain relief by producing increased stimulation of cutaneous mechanoreceptors, and provides muscle activation.

Akbaba et. al. investigated the effects of kinesio tape in management of rotator cuff tear and found that application of KT is effective in improving pain and function but the improvement was not clinically significant . Desjardins et. al. studied the efficacy of KT for rotator cuff tendonitis and found that KT significantly improved pain free range of motion. However, it couldn't be concluded with sufficient evidence that tendonitis was reduced significantly.

ELIGIBILITY:
Inclusion Criteria:

Both Gender / Age b/w 25-60 Shoulder Pain at rest Positive Neer's Test Positive Drop Arm Test Positive Empty Can Test Positive Hawkin's Kennedy Test

Exclusion Criteria:

* Cervical Post op, referred pain, radiculopathy, open wound, allergy to KT

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2018-12-15 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
Visual Analogue scale | change from baseline.This tool is used to measure pain intensity
  Visual analogue scale (VAS) is a psychometric measuring instrument designed to document the characteristics of disease-related symptom severity in individual patients and use this to achieve a rapid (statistically measurable and reproducible) classification of symptom severity and disease control.
Shoulder Pain and Disability Index | change from baseline.This tool is used to measure pain and disability level.
  The Shoulder Pain and Disability Index (SPADI) is a self-administered questionnaire that consists of two dimensions, one for pain and the other for functional activities. The pain dimension consists of five questions regarding the severity of an individual's pain. Functional activities are assessed with eight questions designed to measure the degree of difficulty an individual has with various activities of daily living that require upper-extremity use. The SPADI takes 5 to 10 minutes for a patient to complete and is the only reliable and valid region-specific measure for the shoulder.

SECONDARY OUTCOMES:
Goniometry | change from baseline.This tool is used to measure range of motion of shoulder joint
  Use to measure joint range of motion

CONTACTS AND LOCATIONS:
Overall Officials: imran Amjad, phd*, Principal Investigator — Associate Professor
Locations (1):
- Imran Amjad, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Oliveira FCL, Pairot de Fontenay B, Bouyer LJ, Desmeules F, Roy JS. Effects of kinesiotaping added to a rehabilitation programme for patients with rotator cuff tendinopathy: protocol for a single-blind, randomised controlled trial addressing symptoms, functional limitations and underlying deficits. BMJ Open. 2017 Sep 24;7(9):e017951. doi: 10.1136/bmjopen-2017-017951. PMID 28947462
- [Background] Redondo-Alonso L, Chamorro-Moriana G, Jimenez-Rejano JJ, Lopez-Tarrida P, Ridao-Fernandez C. Relationship between chronic pathologies of the supraspinatus tendon and the long head of the biceps tendon: systematic review. BMC Musculoskelet Disord. 2014 Nov 18;15:377. doi: 10.1186/1471-2474-15-377. PMID 25408141
- [Background] 3. Cubała A, Śniegocki M, Hoffman J, et al. Use of the kinesio taping method in painful shoulder syndrome. Medical and Biological Sciences2012;26:71-6
- [Background] Aguilar-Ferrandiz ME, Castro-Sanchez AM, Mataran-Penarrocha GA, Guisado-Barrilao R, Garcia-Rios MC, Moreno-Lorenzo C. A randomized controlled trial of a mixed Kinesio taping-compression technique on venous symptoms, pain, peripheral venous flow, clinical severity and overall health status in postmenopausal women with chronic venous insufficiency. Clin Rehabil. 2014 Jan;28(1):69-81. doi: 10.1177/0269215512469120. Epub 2013 Feb 20. PMID 23426563
- [Background] Drouin JL, McAlpine CT, Primak KA, Kissel J. The effects of kinesiotape on athletic-based performance outcomes in healthy, active individuals: a literature synthesis. J Can Chiropr Assoc. 2013 Dec;57(4):356-65. PMID 24302784
- [Background] Lin JJ, Hung CJ, Yang PL. The effects of scapular taping on electromyographic muscle activity and proprioception feedback in healthy shoulders. J Orthop Res. 2011 Jan;29(1):53-7. doi: 10.1002/jor.21146. PMID 20607815
- [Background] 7. Akbaba YA, Mutlu EK, Altun S, Gümüşoğlu G, Çelik D. The effects of Kinesio Tape application with different verbal input given to with patients with rotator cuff tear. Orthopaedic Journal of Sports Medicine. 2017;5(2 suppl2):2325967117S00058.
- [Background] Kaya DO, Baltaci G, Toprak U, Atay AO. The clinical and sonographic effects of kinesiotaping and exercise in comparison with manual therapy and exercise for patients with subacromial impingement syndrome: a preliminary trial. J Manipulative Physiol Ther. 2014 Jul-Aug;37(6):422-32. doi: 10.1016/j.jmpt.2014.03.004. Epub 2014 Aug 6. PMID 25108752
- [Background] Kim MH, Oh JS. Effects of humeral head compression taping on the isokinetic strength of the shoulder external rotator muscle in patients with rotator cuff tendinitis. J Phys Ther Sci. 2015 Jan;27(1):121-2. doi: 10.1589/jpts.27.121. Epub 2015 Jan 9. PMID 25642053
- [Background] Senbursa G, Baltaci G, Atay OA. The effectiveness of manual therapy in supraspinatus tendinopathy. Acta Orthop Traumatol Turc. 2011;45(3):162-7. doi: 10.3944/AOTT.2011.2385. PMID 21765229